CLINICAL TRIAL: NCT01203917
Title: An Open Label, Multicentre, Single Arm Study to Characterise the Efficacy, Safety and Tolerability of Gefitinib 250 mg (IRESSA™) as First Line Treatment in Caucasian Patients, Who Have Epidermal Growth Factor Receptor (EGFR) Mutation Positive Locally Advanced or Metastatic Non-Small Cell Lung Cancer
Brief Title: Efficacy, Safety, Tolerability of Gefitinib as 1st Line in Caucasian Patients With EGFR Mutation Positive Advanced NSCLC
Acronym: IFUM
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D791AC00014
Record Dates: First submitted 2010-09-07; First posted 2010-09-17 (Estimated); Results first posted 2013-10-14 (Estimated); Last update posted 2017-01-02 (Estimated); Status verified 2016-11

CONDITIONS: Caucasian Patients With EGFR Mutation Positive Advanced NSCLC
Keywords: Gefitinib; EGFR TKI; efficacy; Caucasian patients; EGFR mutation positive advanced NSCLC; safety
MeSH Terms: interventions — Gefitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Other): gefitinib 250mg tablet
  Interventions: Drug: Gefitinib

INTERVENTIONS:
Drug: Gefitinib — 250mg tablet oral, once daily until objective disease progression is documented or until other discontinuation criterion is met
  Other Names: IRESSA™

SUMMARY:
This study is carried out to see how Caucasian patients with lung cancer which has EGFR mutation will respond to gefitinib (IRESSA™) as a first line treatment. Safety data will also be collected and analysed to confirm that treatment with gefitinib is safe and well tolerated.

DETAILED DESCRIPTION:
An Open Label, Multicentre, Single Arm Study to Characterise the Efficacy, Safety and Tolerability of Gefitinib 250 mg (IRESSA™) as First line Treatment in Caucasian Patients, who have Epidermal Growth Factor Receptor (EGFR) Mutation Positive Locally Advanced or Metastatic Non-Small Cell Lung Cancer

ELIGIBILITY:
Inclusion Criteria:

* Locally advanced or metastatic non-small cell lung cancer (i.e. cancer that has spread from where it started) which is EGFR mutation positive
* Caucasian female or male patients aged 18 years or over
* Measurable disease, i.e. at least one lesion, not previously irradiated, as ≥ 10 mm in the longest diameter (≥ 15 mm in short axis for lymph node )

Exclusion Criteria:

* Prior adjuvant chemotherapy or other systemic anti-cancer treatment less than 6 month, or palliative radiotherapy less than 4 weeks prior to start of study treatment.
* Brain metastases or spinal cord compression, unless treated and stable without steroids
* Any clinically significant illness, which will jeopardize the patients' safety and their participation in the study.

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1060 (Actual)
Dates: Start 2010-09; Primary Completion 2012-08 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Haiyi Jiang, Study Director — AstraZeneca
Locations (61):
- Bulgaria (5):
  - Research Site, Plovdiv
  - Research Site, Sofia
  - Research Site, Stara Zagora
  - Research Site, Varna
  - Research Site, Vratsa
- France (2):
  - Research Site, Angers
  - Research Site, Saint-Herblain
- Greece (4):
  - Research Site, Athens
  - Research Site, Heraklion
  - Research Site, Larissa
  - Research Site, Thessaloniki
- Hungary (6):
  - Research Site, Budapest
  - Research Site, Deszk
  - Research Site, Edelény
  - Research Site, Győr
  - Research Site, Mosdós
  - Research Site, Székesfehérvár
- Italy (4):
  - Research Site, Ancona
  - Research Site, Carpi
  - Research Site, Livorno
  - Research Site, Perugia
- Norway (3):
  - Research Site, Oslo
  - Research Site, Stavanger
  - Research Site, Trondheim
- Poland (9):
  - Research Site, Gdansk
  - Research Site, Krakow
  - Research Site, Lubin
  - Research Site, Olsztyn
  - Research Site, Otwock
  - Research Site, Szczecin
  - Research Site, Torun
  - Research Site, Warsaw
  - Research Site, Wroclaw
- Portugal (4):
  - Research Site, Coimbra
  - Research Site, Lisbon
  - Research Site, Porto
  - Research Site, Vila Nova de Gaia
- Romania (4):
  - Research Site, Brasov
  - Research Site, Bucharest
  - Research Site, Cluj-Napoca
  - Research Site, Constanța
- Spain (5):
  - Research Site, Lleida
  - Research Site, Lugo
  - Research Site, Madrid
  - Research Site, Majadahonda
  - Research Site, Málaga
- Switzerland (4):
  - Research Site, Basel
  - Research Site, Chur
  - Research Site, Rapperswil-Jona
  - Research Site, Sursee
- Turkey (Türkiye) (3):
  - Research Site, Ankara
  - Research Site, Istanbul
  - Research Site, Izmir
- United Kingdom (8):
  - Research Site, Aberdeen
  - Research Site, Birmingham
  - Research Site, Burnley
  - Research Site, Cambridge
  - Research Site, Dundee
  - Research Site, Liverpool
  - Research Site, Nottingham
  - Research Site, Wolverhampton

REFERENCES:
- [Derived] Douillard JY, Ostoros G, Cobo M, Ciuleanu T, McCormack R, Webster A, Milenkova T. First-line gefitinib in Caucasian EGFR mutation-positive NSCLC patients: a phase-IV, open-label, single-arm study. Br J Cancer. 2014 Jan 7;110(1):55-62. doi: 10.1038/bjc.2013.721. Epub 2013 Nov 21. PMID 24263064

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 1060 Caucasian patients with locally advanced or metastatic NSCLC were screened, and 118 patients had activating sensitizing EGFR mutation eligible for the study (EGFR M+). 106 EGFR M+ patients received at least 1 dose of gefitinib. One patient had EGFR mutation not eligible for the study (EGFR M+I) and was started on gefitinib in error.
Groups:
- Gefitinib: Gefitinib 250 mg oral tablets once daily, administered continuously from Visit 2 until objective disease progression was documented or any other criterion for discontinuation was met. Gefitinib tablets were taken at approximately the same time each day.
Period: Overall Study
Arm/Group | Gefitinib
Started | 107 (106 patients were EGFR M+ patients and 1 patient was EGFR M+I)
Completed | 71 (Patients on-going study at data cut-off(of which 49 were still on study treatment).)
Not Completed | 36
Not completed — Death | 29
Not completed — Lost to Follow-up | 2
Not completed — Withdrawal by Subject | 3
Not completed — Due to objective disease progression | 1
Not completed — Due to EGFR M+I patient | 1

BASELINE CHARACTERISTICS:
Population: This is a subset of all the screened patients who are found to be EGFR M+ and who have taken at least one dose of study medication (i.e. EGFR M+ patients are those who have activating sensitising EGFR mutation eligible for the study).
Arm/Group | Gefitinib
Number analyzed (Participants) | 106
Age, Continuous [Mean (Standard Deviation); unit: Years] | 64.0 (11.81)
Age, Customized [Number; unit: Participants]
  > =18 to < 65 Years | 52
  > =65 to < 75 Years | 28
  > =75 Years | 26
Gender [Count of Participants; unit: Participants]
  Female | 75
  Male | 31
Race/Ethnicity, Customized [Number; unit: Participants]
  White | 106
  Other | 0

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR) (Investigator)
Description: % of patients in the Full analysis set who have a complete response [CR] or partial response [PR] confirmed by repeat imaging at least 4 weeks later with no evidence of progression between confirmation visits (as defined by Response Evaluation Criteria in Solid Tumours version 1.1 (RECIST 1.1)). CR: disappearance of all target lesions (TLs) & non-target lesions (NTLs). PR: >= 30% decrease in the sum of diameters compared to baseline (with no evidence of progression) and the NTLs are at least stable with no evidence of new lesions. Outcome is based on measurements made at site by investigator.
Time Frame: Scans taken at baseline and then follow up assessments taken every 6 weeks until progression, or last evaluable assessment in the absence of progression, assessed up to 23 months
Population: Full analysis set, EGFR M+ patients who had taken at least 1 dose of gefitinib
Measure: Number; unit: Percentage of Participants
Arm/Group | Gefitinib
Number analyzed (Participants) | 106
Percentage of Participants
  % Responders | 69.8
  % Non-responders | 30.2

2. Secondary Outcome: Disease Control Rate (DCR) (Investigator)
Description: DCR is calculated as the % of the FAS patient population with a best visit response of CR, PR (a visit response of CR or PR which is confirmed at least 4 weeks later) or stable disease (SD). SD is defined as no evidence of CR, PR or progression and must have occurred at a minimum of 6 weeks after first dose of study treatment. (progression is defined as ≥20% increase in the sum of the diameters of target lesions from minimum; clinically significant progression in non-target lesions; the presence of a new lesion or death). Outcome is based on measurements made at site by investigator.
Time Frame: as for outcome 1
Population: Full analysis set, EGFR M+ patients who had taken at least 1 dose of gefitinib
Measure: Number; unit: Percentage of Participants
Arm/Group | Gefitinib
Number analyzed (Participants) | 106
Percentage of Participants
  % Controlled | 90.6
  % Uncontrolled | 9.4

3. Other Pre Specified Outcome: Disease Control Rate (DCR) (Independent Central Review)
Description: DCR is calculated as the % of the FAS patient population with a best visit response of CR, PR (a visit response of CR or PR which is confirmed at least 4 weeks later) or stable disease (SD). SD is defined as no evidence of CR, PR or progression and must have occurred at a minimum of 6 weeks after first dose of study treatment. (progression is defined as ≥20% increase in the sum of the diameters of target lesions from minimum; clinically significant progression in non-target lesions; the presence of a new lesion or death). Outcome is based on measurements of scans by central review.
Time Frame: as for outcome 1
Population: Full analysis set, EGFR M+ patients who had taken at least 1 dose of gefitinib
Measure: Number; unit: Percentage of Participants
Arm/Group | Gefitinib
Number analyzed (Participants) | 106
Percentage of Participants
  % Controlled | 88.7
  % Uncontrolled | 11.3

4. Other Pre Specified Outcome: Objective Response Rate (ORR) (Independent Central Review))
Description: % of patients in the Full analysis set who have a complete response [CR] or partial response [PR] confirmed by repeat imaging at least 4 weeks later with no evidence of progression between confirmation visits (as defined by Response Evaluation Criteria in Solid Tumours version 1.1 (RECIST 1.1)). CR: disappearance of all target lesions (TLs) & non-target lesions (NTLs). PR: >= 30% decrease in the sum of diameters compared to baseline (with no evidence of progression) and the NTLs are at least stable with no evidence of new lesions. Outcome is based on measurements of scans by central review.
Time Frame: as for outcome 1
Population: Full analysis set, EGFR M+ patients who had taken at least 1 dose of gefitinib
Measure: Number; unit: Percentage of Participants
Arm/Group | Gefitinib
Number analyzed (Participants) | 106
Percentage of Participants
  % Responders | 50.0
  % Non-responders | 50.0

5. Secondary Outcome: Progression - Free Survival (PFS) (Investigator)
Description: PFS was defined as the time from the first dose of gefitinib study treatment until objective disease progression as defined by RECIST 1.1 (≥20% increase in the sum of the diameters of target lesions from minimum, clinically significant progression in non-target lesions or the presence of a new lesion) or death (by any cause in the absence of progression). Progression is based on measurements made at site by investigator.
Time Frame: as for outcome 1
Population: Full analysis set, EGFR M+ patients who had taken at least 1 dose of gefitinib
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Gefitinib
Number analyzed (Participants) | 106
Months | 9.72 [8.48 to 11.04]

6. Other Pre Specified Outcome: Progression - Free Survival (PFS) (Independent Central Review)
Description: PFS was defined as the time from the first dose of gefitinib study treatment until objective disease progression as defined by RECIST 1.1 (≥20% increase in the sum of the diameters of target lesions from minimum, clinically significant progression in non-target lesions or the presence of a new lesion) or death (by any cause in the absence of progression). Progression is based on measurements of scans by central review.
Time Frame: as for outcome 1
Population: Full analysis set, EGFR M+ patients who had taken at least 1 dose of gefitinib
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Gefitinib
Number analyzed (Participants) | 106
Months | 6.97 [6.41 to 9.86]

7. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time from first dose of gefitinib study treatment until death by any cause. Patients who had not died at the time of analysis were censored at the last date the patient was known to be alive.
Time Frame: Survival follow up from first dose of gefitinib till death of the patient or till end of study in absence of death.
Population: Full analysis set, EGFR M+ patients who had taken at least 1 dose of gefitinib
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Gefitinib
Number analyzed (Participants) | 106
Months | 19.22 [16.95 to NA] — The upper limit of 95% Confidence interval for Overall Survival was longer than 19.22 and was not observed during the trial period.

ADVERSE EVENTS:
Arm/Group | Gefitinib 250 mg
Serious Adverse Events (participants affected / at risk) | 21/107
Other Adverse Events (participants affected / at risk) | 87/107
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gefitinib 250 mg (N=107)
ANAEMIA (Blood and lymphatic system disorders) | 1 (1)
CARDIAC FAILURE (Cardiac disorders) | 2 (3)
VERTIGO (Ear and labyrinth disorders) | 1 (1)
DIARRHOEA (Gastrointestinal disorders) | 2 (2)
VOMITING (Gastrointestinal disorders) | 3 (3)
ASTHENIA (General disorders) | 1 (1)
GASTROENTERITIS (Infections and infestations) | 1 (1)
PNEUMONIA (Infections and infestations) | 3 (3)
POSTOPERATIVE WOUND INFECTION (Infections and infestations) | 1 (1)
VIRAL INFECTION (Infections and infestations) | 1 (1)
ANKLE FRACTURE (Injury, poisoning and procedural complications) | 1 (1)
FEMORAL NECK FRACTURE (Injury, poisoning and procedural complications) | 1 (1)
RADIUS FRACTURE (Injury, poisoning and procedural complications) | 1 (1)
TIBIA FRACTURE (Injury, poisoning and procedural complications) | 1 (1)
DECREASED APPETITE (Metabolism and nutrition disorders) | 1 (1)
DEMENTIA ALZHEIMER'S TYPE (Nervous system disorders) | 1 (1)
HYPOAESTHESIA (Nervous system disorders) | 1 (1)
SENILE DEMENTIA (Nervous system disorders) | 1 (1)
TRANSIENT ISCHAEMIC ATTACK (Nervous system disorders) | 1 (1)
HAEMOPTYSIS (Respiratory, thoracic and mediastinal disorders) | 1 (1)
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 2 (2)
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 1 (1)
SKIN NECROSIS (Skin and subcutaneous tissue disorders) | 1 (1)
HYPERTENSION (Vascular disorders) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gefitinib 250 mg (N=107)
DIARRHOEA (Gastrointestinal disorders) | 31 (55)
NAUSEA (Gastrointestinal disorders) | 11 (14)
VOMITING (Gastrointestinal disorders) | 12 (13)
ASTHENIA (General disorders) | 12 (12)
URINARY TRACT INFECTION (Infections and infestations) | 7 (10)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 9 (10)
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 7 (8)
DECREASED APPETITE (Metabolism and nutrition disorders) | 10 (11)
HEADACHE (Nervous system disorders) | 6 (6)
COUGH (Respiratory, thoracic and mediastinal disorders) | 12 (12)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 7 (7)
DERMATITIS ACNEIFORM (Skin and subcutaneous tissue disorders) | 7 (7)
DRY SKIN (Skin and subcutaneous tissue disorders) | 12 (13)
RASH (Skin and subcutaneous tissue disorders) | 50 (65)
HYPERTENSION (Vascular disorders) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less